CLINICAL TRIAL: NCT06231940
Title: Experimental Study on the Efficacy of Complex Decongestive Therapy (CDT) Treatment in Patients With Venous Insufficiency
Brief Title: Efficacy of Complex Decongestive Therapy (CDT) in Patients With Venous Insufficiency: a Experimental Study
Acronym: CDT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Beatriz-María Bermejo-Gil, Principal Investigator, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CDT-USAL
Record Dates: First submitted 2024-01-08; First posted 2024-01-30 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Lymphatic Edema; Cellulitis of Leg; Vein Disease
Keywords: conservative treatment; Venous Insufficiency; Complex decongestive therapy
MeSH Terms: conditions — Lymphedema; Venous Insufficiency | interventions — carbohydrate-deficient transferrin

STUDY DESIGN:
Intervention Model Description: The experimental group undergoes twice-weekly CDT sessions, including manual lymph drainage, pneumatic compression, and bandaging, while the control group receives no treatment.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Complex Decongestive Therapy (CDT) in venous insufficiency (Experimental)
  Interventions: Other: Complex Decongestive Therapy (CDT) in venous insufficiency,
- Control group (No Intervention)

INTERVENTIONS:
Other: Complex Decongestive Therapy (CDT) in venous insufficiency, — Complex Decongestive Therapy (CDT) is a comprehensive treatment approach primarily used for lymphedema and related conditions, but it's also beneficial for chronic venous insufficiency and other edematous conditions. CDT aims to reduce swelling and maintain the reduction, improve skin condition, and alleviate symptoms. It typically involves two phases: an intensive phase to reduce swelling as much as possible and a maintenance phase to sustain the achieved results. The main components of CDT include: Manual Lymph Drainage (MLD),Compression Therapy, Exercise, Skin Care, Education and Self-Care:
  Arms: Complex Decongestive Therapy (CDT) in venous insufficiency

SUMMARY:
The study investigates the effectiveness of Complex Decongestive Therapy (CDT) in improving venous flow and reducing symptoms in venous insufficiency patients. The primary goal is to demonstrate CDT's effects, with secondary goals assessing symptom relief, life quality improvement, and adverse effects. The trial is a simple blind randomized design, involving an experimental group receiving CDT plus exercises and a control group doing exercises alone. Participants are adults with specific classifications of venous insufficiency, excluding certain health conditions. The study will involve 12 participants in the experimental group and 9 in the control group.

DETAILED DESCRIPTION:
The study hypothesizes that Complex Decongestive Therapy (CDT) is effective in increasing venous flow and reducing symptoms in patients with venous insufficiency. The primary objective is to demonstrate the effects of CDT in these patients. Secondary objectives include evaluating if physiotherapy treatment increases venous flow, decreases symptoms (edema, pain, heaviness, and fatigue), and improves patient quality of life, assessing adverse effects post-intervention, determining the reliability of circumferential edema measurement, and correlating venous insufficiency with various risk factors and aggravating conditions.

The design is a simple blind randomized clinical trial comparing an experimental group receiving CDT and lower limb exercise program to a control group doing standardized preventive measures. Participants include both men and women over 18 years old with clinical classification of C2-C5 venous insufficiency, excluding those with specific acute or unmanaged chronic conditions, or those currently or recently treated with CDT. The experimental group consists of 12 participants receiving CDT and exercise, while the control group includes 9 participants following the exercise program.

The study focuses on various variables to assess the effectiveness of Complex Decongestive Therapy (CDT) in patients with venous insufficiency, including venous reflux, flow and diameter of specific veins, intracellular and extracellular fluid volumes, and edema measurements at different lower limb sites. It also evaluates symptom severity and quality of life using validated questionnaires (CEAP, VCSS, CIVIQ-20).

Measurement tools include ultrasound for venous flow and diameter, bioimpedance for cellular fluids, and a tape measure for limb circumference. Assessments will be done using ultrasound and physiotherapy evaluations, along with patient-completed questionnaires.

The intervention involves pre and post-intensive 4-week CDT treatment evaluations, with a follow-up one month later. The experimental group undergoes twice-weekly CDT sessions, including manual lymph drainage, pneumatic compression, and bandaging, while the control group receives no treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 35 and 75 years
* Presence of mild venous insufficiency, moderate or severe (grades C1, C2, C3, and C4 on the Clinical, Etiologic, Anatomic, Pathophysiologic [CEAP] scale).

Exclusion Criteria:

* Subjects affected by uncompensated acute cardiac, hepatic, and renal disease, acute obstructive vascular disease, acute trauma, primary lymphedema, and acute skin infections.
* Patients who are currently receiving complex decongestive therapy treatment or in the last six months.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — self-identified gender will be included and gender identity question will be ask to analyze gender-diverse related to health correlations
Enrollment: 21 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Vein flow | pre-intervention and immediately after the intervention
  vein flow by echograph
Internal saphenous vein diameter | pre-intervention and immediately after the intervention
  vein flow by echograph
intracellular and extracellular fluid in each of the lower extremities | pre-intervention and immediately after the intervention
  Bioimpedance meter for intracellular and extracellular segmental fluid measurement
lower extremities edema | pre-intervention and immediately after the intervention
  Measuring tape for limb circumference measurement
venous insufficiency involvement | pre-intervention and immediately after the intervention
  CEAP questionnaire (Clinical, Etiologic, Anatomic, and Pathophysiologic).CEAP Classification for Chronic Venous Disorders. Ranges from C0 to C6. The minimum on the clinical scale is C0 (no signs of venous disease). The maximum is C6 (active venous ulcer).
severity of venous insufficiency | pre-intervention and immediately after the intervention
  Venous Clinical Severity Score (VCSS). Includes 9 clinical categories, each scored from 0-3. Minimum score 0 (no symptoms or signs). Mazimum score 27 (the wors severy, severe venous disease)
Perceived Quality of Life | pre-intervention and after the intervention
  Chronic Venous Insufficiency Questionnaire-20 (CIVIQ-20). It consists on 20 questions scored on5-point likert scale. Minimum score 20 (best possible quality of life, leas impact of venous insufficiency) maximum score 100 (worst quality of life)

CONTACTS AND LOCATIONS:
Locations (1):
- Beatriz María Bermejo Gil, Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF